CLINICAL TRIAL: NCT04350151
Title: National French Survey on Psychological Distress at Work of Anesthesia and Intensive Care Residents
Acronym: PSY-DESAR
Status: Completed | Type: Observational
Sponsor: Facteurs Humains en Santé (Other)
Collaborators: Dominique FLETCHER MD-PhD (Unknown); François Marty MD (Unknown); Dinh Phong Nguyen MD (Unknown); Loic Druette MD (Unknown); Benoit Plaud MD-PhD (Unknown); Clément Duret MD (Unknown)
Responsible Party: Principal Investigator, François JAULIN, Principal Investigator, Facteurs Humains en Santé
Other Study IDs: 20200316
Record Dates: First submitted 2020-03-16; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Burnout, Professional; Intensive Care; Anesthesia; Depression, Anxiety; Stress, Psychological; Fatigue; Work Load
MeSH Terms: conditions — Burnout, Professional; Depression; Anxiety Disorders; Stress, Psychological; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: no intervention — no intervention

SUMMARY:
Psychological distress is a significant problem for healthcare professionals and students in training. The investigator question the prevalence of this problem in French residents in anaesthesia and intensive care training.

DETAILED DESCRIPTION:
The investigator performed an observational study on the national population of anaesthesia residents. A questionnaire was sent to all residents composed with validated questionnaires analyzing psychological distress (Hospital Anxiety and Depression Scale (HADS), Copenhagen Burnout Inventory (CBI), Perceived Stress Scale (PSS), Karasek's questionnaire; work-related questions (work hours per week, night shift per month, application of safety rest after night shift, average time to start and end work, break time and time for food per day; two semi-open work-related questions (main stressor during internship, professional orientation); a free verbatim.

ELIGIBILITY:
Inclusion Criteria:

* resident of intensive care or anesthesia, french

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: French resident of intensive care and anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | baseline
  Investigation of the anxiety and depression with 14 questions, the cut-off score is more than 11 for anxiety or depression
Copenhagen Burnout Inventory (CBI) | baseline
  Investigation of the burnout on 3 axes: personal, professional and relational with 19 questions, the cut-off score is 50 to identify a burnout
Karacek's questionnaire | baseline
  Investigation of the stress at work
Perceived Stress Scale (PSS) | baseline
  Investigation of the stress with 10 questions

OTHER OUTCOMES:
Workload | baseline
  number of work-hours per week
Gender | baseline
  Male, female

CONTACTS AND LOCATIONS:
Locations (1):
- Facteurs Humains en Santé, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
At the end of the survey
Supporting Information: Study Protocol, SAP, CSR